CLINICAL TRIAL: NCT05321355
Title: Study on Disease Course and Quality of Life in Patients With Sleep Disorders (Mainz Sleep Registry)
Brief Title: Mainz Register of Patients With Sleep Disorders
Acronym: MAINZ-SLEEPREG
Status: Recruiting | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Dr. Yaroslav Winter, Head of Mainz Comprehensive Epilepsy and Sleep Medicine Center, Johannes Gutenberg University Mainz
Other Study IDs: MAINZ-SLEEPREG
Record Dates: First submitted 2022-04-04; First posted 2022-04-11 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Sleep Disorder; Sleep Disorder Parasomnia; Narcolepsy; Sleep Apnea; Insomnia; Somnambulism; Idiopathic Hypersomnia; Restless Legs Syndrome; REM Behavior Disorder
MeSH Terms: conditions — Sleep Wake Disorders; Parasomnias; Narcolepsy; Sleep Apnea Syndromes; Sleep Initiation and Maintenance Disorders; Somnambulism; Idiopathic Hypersomnia; Restless Legs Syndrome; REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with narcolepsy treated with vagus nerve stimulation: Patient with narcolepsy treated with vagus nerve stimulation
  Interventions: Device: Implantation of vagus nerve stimulation according to clinical indication
- Patient without narcolepsy treated with vagus nerve stimulation: Patient without narcolepsy treated with vagus nerve stimulation
  Interventions: Device: Implantation of vagus nerve stimulation according to clinical indication

INTERVENTIONS:
Device: Implantation of vagus nerve stimulation according to clinical indication — no interventions, only observation

SUMMARY:
Prospective longitudinal observational registry study of all patients with sleep disorders treated in the Mainz Comprehensive Epilepsy and Sleep Medicine Center with the focus on the course of the disease and quality of life.

DETAILED DESCRIPTION:
Clinical parameters of patients, such as onset of the disease, prior medication, disease severity, which are important for the data analysis also collected retrospectively before the initiation of the registry. Data on the quality of life is collected only prospectively

ELIGIBILITY:
Inclusion Criteria:

* patients with narcolepsy
* patients with other neurological sleep disorders

Exclusion Criteria:

* patients aged <18 years
* patients who cannot provide informed consent and don't have a legal guardian

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated in Mainz Comprehensive Epilepsy and Sleep Medicine Center
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Excessive daytime sleepiness (EDS) as measure by Epworth Sleepiness Scale (ESS) after 3 months (rating from 0 (no sleepiness) to 24 (severe sleepiness)) | 3 months
  EDS measure by ESS at the follow-up after 3 months
European Quality of Life 5 dimensions Index (EQ 5D Index) | 3 months
  health-related quality of life measured by EQ5D-Index (European Quality of Life 5 dimensions), rating from 0 (worst possible state) to 1 (best possible state)
Excessive daytime sleepiness (EDS) as measure by Epworth Sleepiness Scale (ESS) after 6 months | 6 months
  EDS measure by ESS at the follow-up after 6 months (rating from 0 (no sleepiness) to 24 (severe sleepiness))
European Quality of Life 5 dimensions Index (EQ 5D Index) | 6 months
  health-related quality of life measured by EQ5D-Index (European Quality of Life 5 dimensions), rating from 0 (worst possible state) to 1 (best possible state)

SECONDARY OUTCOMES:
Multidimensional Fatigue Inventory | 3 months
  Multidimensional Fatigue Inventory: 20-item self-report instrument designed to measure fatigue. Measures range from 0-100, representing more severe fatigue at higher scores
Multidimensional Fatigue Inventory | 6 months
  Multidimensional Fatigue Inventory: 20-item self-report instrument designed to measure fatigue. Measures range from 0-100, representing more severe fatigue at higher scores
Beck Depression Inventory II | 6 months
  Beck Depression Inventory II: higher scores correspond to more severe depression (range 0-63)
Beck Depression Inventory II | 12 months
  Beck Depression Inventory II: higher scores correspond to more severe depression (range
Resilience Scale 13 | 6 months
  Resilience Scale 13 (short version with 13 questions): 13-66 points correspond with low resilience, 67-72 with moderate and 73-91 with high resilience
Resilience Scale 13 | 12 months
  Resilience Scale 13 (short version with 13 questions): 13-66 points correspond with low
European Quality of Life visual analogue scale (EQ-VAS) | 6 months
  European Quality of Life visual analogue scale (EQ-VAS) (ranges from 0 to 100, where 0 is the worst anf 100 the best state)
European Quality of Life visual analogue scale (EQ-VAS) | 12 months
  European Quality of Life visual analogue scale (EQ-VAS) (ranges from 0 to 100, where 0 is the worst anf 100 the best state)
Ullanlinna Narcolepsy Scale (UNS) | 3 months
  scale to identify the burden of narcolepsy
Ullanlinna Narcolepsy Scale (UNS) | 6 months
  scale to identify the burden of narcolepsy
World Health Organization Quality of Life-BREF (WHOQOL-BREF) | 6 months
  World Health Organization Quality of Life-BREF (WHOQOL-BREF), a scale to assess overall quality of life with a range 0-100 (higher scores correspond better quality of life)
World Health Organization Quality of Life-BREF (WHOQOL-BREF) | 12 months
  World Health Organization Quality of Life-BREF (WHOQOL-BREF), a scale to assess overall quality of life with a range 0-100 (higher scores correspond better quality of life)
Pittsburgh Sleep Quality Index | 6 months
  Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances, scoring between 0 and 21 with higher scores corresponding to worse sleep quality
Pittsburgh Sleep Quality Index | 12 months
  Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances, scoring between 0 and 21 with higher scores corresponding to worse sleep quality
Berlin Social Support Scales (BSSS) | 6 months
  Berlin Social Support Scales (BSSS) is used to assess the amount of emotional, informational and instrumental support received by patients: Total scores ranged from 15 to 60, higher scores identify better support
Berlin Social Support Scales (BSSS) | 12 months
  Berlin Social Support Scales (BSSS) is used to assess the amount of emotional, informational and instrumental support received by patients: Total scores ranged from 15 to 60, higher scores identify better support

CONTACTS AND LOCATIONS:
Locations (1):
- Mainz Comprehensive Epilepsy and Sleep Medicine Center, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Winter Y, Lang C, Kallweit U, Apel D, Fleischer V, Ellwardt E, Groppa S. Pitolisant-supported bridging during drug holidays to deal with tolerance to modafinil in patients with narcolepsy. Sleep Med. 2023 Dec;112:116-121. doi: 10.1016/j.sleep.2023.10.005. Epub 2023 Oct 9. PMID 37839272